CLINICAL TRIAL: NCT00469534
Title: A Pilot Study Evaluating Minimized Time to Beam Hypofractionated IMRT With PET-Assisted Target Definition in Patients With High Grade Gliomas
Brief Title: Minimized Time to Beam in Patients With High Grade Gliomas
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-9-0039
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: High Grade Glioma
Keywords: minimized time to beam; hypofractionated 3D CRT plus IMRT; PET-scan
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: IMRT

SUMMARY:
A Pilot Study Evaluating Minimized Time to Beam Hypofractionated IMRT with PET Assisted Target Definition in Patients with High Grade Gliomas

The aim of this pilot project is to explore the feasibility of combining a simple conformal plan (Phase I) with an IMRT treatment approach (Phase II) for high grade glioma patients with the aim of starting the RT as soon as possible following the patient's first outpatient visit (thus, minimized 'time to beam'). It is hoped that the rapid treatment start with the initial 3D CRT plan will lessen clinical deterioration due to the growth of these aggressive tumours. The use of Linac-based IMRT in Phase II of the patient's treatment plan will maintain the benefit of the sophistication of IMRT.

Using novel PET imaging we also hope to better characterize regions of glioma cells thus producing more optimized planning target volumes (PTVs) for each patient and decreasing the volume of normal brain irradiated with the aim of minimizing radiation toxicities. Hopefully this planning and treatment approach will provide an improvement in the quality of life and outcome for high grade glioma patients.

DETAILED DESCRIPTION:
A Pilot Study Evaluating Minimized Time to Beam Hypofractionated IMRT with PET Assisted Target Definition in Patients with High Grade Gliomas

BACKGROUND INFORMATION Standard Treatment High grade gliomas (HGG) comprise the vast majority of primary brain tumors. With conventional treatment, tumor recurrence and subsequent patient death is expected in all but a small minority of patients. Conventional treatment consists of maximal surgical debulking followed by radiation therapy (RT) and temozolomide (TMZ) chemotherapy. Typically the radiation therapy is given in 2 Gy fractions to a total dose of 60 Gy to the planning target volume (PTV).

What is the Optimal PTV? Currently it is not know what target volume constitutes the optimal PTV for an individual patient with a HGG. With conventional MRI-based target definition, a common practice is to draw a gross tumour volume (GTV) to include the contrast enhancing lesion seen on T1C images. An additional uniform margin of approximately 1.5 cm is added to address clinically occult glioma cells and create the clinical target volume (CTV), plus an additional 0.5 cm to create the final PTV. This practice is based on pattern of recurrence studies. In these studies, 80-90% of the HGGs tended to recur within 2 cm of the original T1C enhancing lesion. The addition of a uniform 2 cm margin to the initial GTV dramatically increases the volume of apparently normal brain irradiated, and the volume of brain irradiated is a principal determinant of subsequent radiation toxicity. By using positron emission tomography (PET) imaging to better characterize which regions harbour glioma cells, we hope to be able to minimize the size of the uniform margins applied to the GTV, and thus produce a more optimized PTV for each patient.

PET Imaging For this pilot study we will be using novel PET agents including F19AZA and C11 Methionine to assist in the construction of a more patient optimized PTV. The volumes constructed based on MRI reflect the underlying anatomy or structure of the tumor. On the other hand the volumes constructed base on PET imaging reflect the underlying physiology and thus will be referred to as the biological target volume (BTV) to distinguish it from the MRI base GTV. The clinician will then use the complementary information provided by the GTV and BTV to construct a composite CTV, and this will be grown with a uniform 0.5 cm margin into the PTV. The PET imaging will be carried out under a separate research protocol submitted by nuclear medicine, and the patient will need to sign an informed consent for each agent used. At the investigators discretion, the patient will be given the choice to undergo imaging using the full complement of PET agents or a selected subset of these agents.

IMRT 3D conformal RT (3D CRT) is the standard treatment technique used to treat HGGs at many centres. With the advancement of IMRT techniques, clinicians are able to deliver more sophisticated RT plans. With these more sophisticated approaches clinicians should be able limit the volume of apparently uninvolved brain encompassed in the high dose treatment volume. In our recent protocol we gained experience using helical tomotherapy-base IMRT. In the current protocol, we plan to use Linac-based IMRT. One of the advantages of Linac-based IMRT over helical tomotherapy is that the plan may include non-coplanar beams. This additional degree of freedom is expected to result in better plan conformation. Also, Linac-based IMRT plans can be added to the conformal plan of phase I and thereby adjusted accordingly.

Overcoming Radio-Resistant Tumor Clonogens In this protocol we plan to use hypofractionated RT (60 Gy in 20 fractions over 4 weeks). Hypofractionation has the advantage of shortening the overall treatment time (which minimizes the opportunity for tumor repopulation during the treatment course). The larger dose per fraction is also expected to be more biologically effective against radio-resistant tumor clonogens. An identical fractionation scheme was reported to be safe in a recent study of patients with HGG (IJROBP 58 1 247-252 2004 Sultanem) and a similar fractions scheme was used in our recent glioma protocol 60 Gy in 22 fractions over 4.5 weeks). As of yet, we have not observed any obvious increased toxicity in these patients (Personal Observation).

Minimizing Time to Beam HGGs are locally aggressive and rapidly growing tumors. The typical presenting symptoms are usually related to the mass effect of the tumor on the adjacent and distant nerve cells. Once the intracranial pressure (ICP) has begun to rise, any subsequent growth of the tumor within the confined space of the skull results in a dramatic increase in ICP and subsequent neuron damage (usually permanent). Hence it is imperative that the initiation of therapy not be delayed. Unfortunately the design of sophisticated IMRT plans base on advanced imaging technology is a complex and potentially time consuming process. When treatment is delayed as a consequence of this process, the patient frequent deteriorates clinically possibly resulting in a permanent decline in quality of life, a decision to discontinue RT or even death. In this protocol we plan to explore the feasibility of a combined approach using 3D CRT and IMRT. The first half of the treatment (2 weeks) will be given using a simple 3D CRT approach based on the patient's preoperative MRI images. This will have the advantage of facilitating a rapid start of RT and hopefully arrest any evolving clinical deterioration which may have occurred (minimizing the time to beam). The goal will be to start the RT as soon as possible from the first OPD visit. The planning, evaluation and QA of the IMRT plan will progress while the patient is undergoing phase I of the treatment.

OBJECTIVES

Primary End Point:

1. Time from initial OPD visit to start of RT compared with historical controls receiving helical tomotherapy base IMRT (Time to Beam)

Secondary End Points:

1. Overall Survival
2. Disease-free survival
3. Patterns of recurrence
4. Toxicity
5. Quality of life
6. Number of patients who complete treatment

STUDY DESIGN

Schema Radiation Therapy Phase I 30 Gy in 10 fractions to PTV1 Using 3D CRT

GTV1 = Intra and peri-tumoural edema seen on preoperative MRI CTV1 = GTV1 + 1.5 cm margin PTV1 = CTV1 + 0.5 cm margin

Note: The 1.5 cm margin added to create the CTV1 may be reduced at the discretion of the clinician in areas of anatomical barriers to glioma spread (i.e. skull, tentorium, etc.)

Phase II 30 Gy in 10 fractions to > 90% of the PTV2

GTV2 = Contrast enhancing lesion BTV = Extent of tumor seen on PET imaging CTV2 = (Union of GTV2 and BTV) + >0.5 cm margin PTV2 = CTV2 + 0.5 cm margin

Note: The margin added to the CTV2 may be enlarged at the discretion of the clinician to a maximum of 1.5 cm. The dose received by the PTV2 regions which encroach within 3 mm, or overlap, a dose limiting critical structure should be restricted to the dose constraints allowed for that particular critical structure. Exceptions may be made at the clinician's discretion when the dose limiting critical structure is grossly involved by tumor.

Chemotherapy Patients will also be offered standard TMZ chemotherapy, but patients who refuse TMZ or are unable to tolerate/receive it, may still enroll in the study.

PET Imaging Studies will be done at baseline and post RT (0, 2, 4, 6, and 12 months).

INCLUSION CRITERIA Histopathologically-confirmed grade III or grade IV supratentorial glioma Age > 18 KPS > 70 No prior radiation therapy to the brain No active prior malignancy Signed study-specific consent form

EXCLUSION CRITERIA No histopathologically-confirmation of grade III or grade IV supratentorial glioma Age < 18 KPS < 70 Prior radiation therapy to the brain Active prior malignancy

RECRUITMENT Number of patients 25 (High Grade Glioma)

STATISTICAL ANALYSIS This is a pilot study comprising a total of 25 high grade glioma patients.

STOPPING RULES Both acute and late toxicities will be of interest in this study as well as disease-free survival, patterns of recurrence and quality of life assessments. Patients will be closely followed by their treating Radiation Oncologist and / or the Research Nurse and any sever adverse events will be reported to the Principal Investigator and the Research Ethics Board as per the set REB guidelines.

DATA SAFETY MONITORING COMMITTEE Any serious adverse event that occurs from the time the consented patient has begun study treatment until 30 days after the end of study treatment must be reported to the participating institution's Research Ethics Board within their REB set reporting guidelines. Any SAE that occurs after the one month post study treatment timeframe that is felt to be related to the study treatment must be reported to the participating institution's Research Ethics Board within the REB set reporting guidelines. If a death is related to study treatment, the REB should receive notification within 24 hours of the event, with a full report to follow. All deaths that occur during a study or within 30 days after last study treatment, regardless of the relationship to the treatment, need to be reported to the REB. A research nurse and / or a radiation oncologist will be responsible for regular monitoring of patients on study treatment. If the number of events meets the stopping criteria listed in point 12.0, accrual will be halted and the Principal Investigator will inform the Research Ethics Board in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* histopathologically-confirmed high grade glioma
* 18+ years of age
* no prior radiation therapy to the brain
* no active prior malignancy
* KPS greater or equal to 70
* singed study-specific consent form

Exclusion Criteria:

* no histopathologically confirmation of high grade glioma
* less than 18 years of age
* prior radiation therapy to the brain
* active prior malignancy
* KPS less than 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Time from initial OPD visit to start of RT compared with historical controls receiving helical tomotherapy base IMRT (Time to Beam).

SECONDARY OUTCOMES:
Overall survival, disease-free survival, patterns of recurrence, toxicity, quality of life, number of patients who complete treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Murtha, MD, Principal Investigator — AHS Cancer Control Alberta